CLINICAL TRIAL: NCT03646903
Title: Reducing Help-Seeking Stigma in Young Adults at Elevated Suicide Risk: A Randomized Controlled Trial
Brief Title: Reducing Help-Seeking Stigma in Young Adults at Elevated Suicide Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Ian Stanley, Research Faculty, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRG-0-141-17
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Suicide; Help-Seeking Behavior; Health Behavior
MeSH Terms: conditions — Suicide; Help-Seeking Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Bias Modification for Help-Seeking Stigma (CBM-HS) (Experimental): CBM-HS is a 15-minute web-based intervention designed to alter maladaptive cognitions related to mental health help-seeking. In this task, individuals are presented with a series of statements regarding beliefs about using mental health services (e.g., "Seeking help for my problems means I am weak"). Individuals then select "True" or "False" in response to each statement. Incorrect responses (i.e., demonstrating help-seeking stigma) are followed by corrective feedback. Conversely, correct responses (i.e., promoting help-seeking) are positively reinforced (e.g., "That's right! You are correct!"). Participants in this condition will complete three separate 15-minute CBM-HS sessions.
  Interventions: Behavioral: Cognitive Bias Modification
- Placebo Cognitive Bias Modification (Placebo Comparator): Participants randomized to this condition will complete a similar CBM task with neutral stimuli. The duration of the CBM-Placebo task will be comparable to the duration of the CBM-HS task (i.e., three 15-minute sessions).
  Interventions: Behavioral: Cognitive Bias Modification
- Self-Directed Psychoeducation (Active Comparator): Participants randomized to this condition will review psychoeducation on mental health literacy, mental illness stigma, and treatment options. Readings will be compiled from resources available in the public domain. The duration of self-directed psychoeducation will be comparable to the duration of study tasks for individuals in the CBM-HS study condition (i.e., three 15-minute sessions).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — Cognitive bias modification (CBM) interventions typically involve the completion of brief, web-based tasks in which individuals are presented with a series of stimuli (e.g., words, sentences) and trained to respond in a manner that is positive or neutral, rather than negative and unhelpful. CBM interventions rely on the premise that repeated reinforcement of adaptive cognitions and a reshaping of negative cognitions enhance functioning and reduce distress.
  Arms: Cognitive Bias Modification for Help-Seeking Stigma (CBM-HS); Placebo Cognitive Bias Modification
Behavioral: Psychoeducation — Psychoeducation-based interventions rely on the premise that enhancing knowledge about psychiatric symptoms and treatment will facilitate treatment engagement.
  Arms: Self-Directed Psychoeducation

SUMMARY:
Although there exist interventions that therapeutically impact suicide risk, the connection of individuals at elevated suicide risk to mental health care services remains an ongoing challenge. One persistent barrier to mental health service utilization is help-seeking stigma-that is, having negative beliefs about the implications of seeking help for mental health problems (e.g., "Seeking help means that I am weak"). Thus, to enhance mental health service use among at-risk individuals, efforts are needed to target help-seeking stigma. Preliminary data from our research group indicate that a novel computerized intervention based on cognitive therapy principles can demonstrably reduce help-seeking stigma and increase connection to care among young adults with untreated psychiatric disorders. However, this intervention has not been tested among individuals who are currently experiencing suicidal ideation and are not engaged in mental health treatment. Testing the efficacy of this computerized intervention among young adults at increased risk for suicide is necessary to address the unique challenge of linking at-risk individuals to potentially life-saving treatments. To this end, this study aims to test the efficacy of a brief web-based intervention, cognitive bias modification for help-seeking stigma (CBM-HS), designed to increase mental health help-seeking intentions and behaviors. A total of 78 young adults with current suicidal ideation who are not currently in treatment and who report elevated levels of help-seeking stigma will be randomly assigned to one of three conditions: (1) CBM-HS; (2) CBM-Placebo (i.e., a sham CBM condition analogous to a placebo pill in a pharmaceutical trial); or (3) psychoeducation. Participants will complete assessments at baseline, mid-intervention, post-intervention, and 2-month follow-up to determine the efficacy of CBM-HS in: (a) modifying stigma-related cognitions around mental health help-seeking and service use and (b) increasing treatment initiation and engagement. Moreover, we will test if reductions in stigma-related cognitions mediate the relationship between study condition and subsequent help-seeking behaviors. Findings from the proposed pilot randomized controlled trial have the potential to enhance connection to care among young adults at elevated suicide risk. Importantly, the brief, web-based nature of the intervention enhances its acceptability, feasibility, and scalability. Should CBM-HS demonstrate efficacy in reducing help-seeking stigma and enhancing connection to care among at-risk individuals, it has the potential to serve as a useful tool in suicide prevention efforts.

ELIGIBILITY:
Inclusion Criteria:

* Current undergraduate student
* Current suicidal ideation (DSI-SS Total Score >0)
* Elevated help-seeking stigma (SSOSH Total Score >24)
* No current mental health service use (i.e., ongoing care with a provider to receive psychiatric medications, therapy, and/or counseling)

Exclusion Criteria:

* Lack of Internet access via a privately-located laptop or desktop computer
* Completing last semester of undergraduate coursework
* Imminent suicide risk (i.e., suicide risk warranting hospitalization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stigma and Barriers to Care for Psychological Problems Scale (PS) | 2-Month Follow-Up
  The 11-item Perceived Stigma and Barriers to Care for Psychological Problems Scale (PS) measures the extent to which various concerns might affect an individual's decision to seek psychiatric treatment. Items are rated on a 5-point scale; scores are summed and higher scores (range: 11-55) indicate greater perceived barriers to care. Individual PS items will also be evaluated consistent with past research.
Self-Stigma of Seeking Help (SSOSH) | 2-Month Follow-Up
  The Self-Stigma of Seeking Help (SSOSH) is a 10-item measure of help-seeking stigma. Responses are rated on a 5-point scale; higher scores (range: 0-50) reflect greater self-stigma.
World Mental Health Composite International Diagnostic Interview (WMH-CIDI) | 2-Month Follow-Up
  The self-report version of the World Mental Health Composite International Diagnostic Interview (WMH-CIDI) Services subscale will be utilized to assess structural and attitudinal barriers to care. Items are evaluated individually and higher scores indicate greater structural and attitudinal barriers to care.
Readiness to Change Scale | 2-Month Follow-Up
  An adaptation of the Readiness to Change Scale will assess readiness to engage in help-seeking behaviors. Responses to each of the 6 items are anchored on an 11-point scale, with higher scores indicating greater readiness to engage in mental health treatment.
Mental Health Treatment Survey | 2-Month Follow-Up
  An adapted version of SAMHSA's National Survey on Drug Use and Health (NSDUH) will be used to assess help-seeking behaviors and mental health service use for general mental health problems and/or suicide-related reasons, specifically.
Intervention Acceptability and Feasibility Questionnaire | 2-Month Follow-Up
  An investigator-developed questionnaire will be administered to determine the acceptability and feasibility of the proposed intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ian H Stanley, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No